CLINICAL TRIAL: NCT07048938
Title: Clinical Effect and Mechanism Study of Five Elements Music Therapy(FEMT) on Depression Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-100R
Record Dates: First submitted 2025-06-12; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Depression Disorder; Depression Disorders; Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Antidepressive Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Five-Element Music 1 Primarily in Gong and Zhi modes combined with antidepressant medication (Experimental)
  Interventions: Combination Product: Five-Element Music 1 combined with antidepressant medication
- Five-Element Music 2 Primarily in Shang and Yu modes combined with antidepressant medication (Active Comparator)
  Interventions: Combination Product: Five-Element Music 2 combined with antidepressant medication
- health control (Other)
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Combination Product: Five-Element Music 1 combined with antidepressant medication — The self-composed musical piece Five Elements Music 1 was selected to intervene with the patients, with the songs primarily based on the Gong tone and Zhi tone in traditional Chinese music. On this basis, the intervention was combined with fluoxetine hydrochloride treatment
  Arms: Five-Element Music 1 Primarily in Gong and Zhi modes combined with antidepressant medication
Combination Product: Five-Element Music 2 combined with antidepressant medication — The self-composed musical piece Five Elements Music 2 was selected to intervene with the patients, with the songs primarily based on the Shang mode (A) and Yu (E) mode in traditional Chinese music. On this basis, the intervention was combined with fluoxetine hydrochloride treatment
  Arms: Five-Element Music 2 Primarily in Shang and Yu modes combined with antidepressant medication
Other: No Intervention: Observational Cohort — No intervention will be applied to healthy people
  Arms: health control

SUMMARY:
The goal of this clinical trial is to learn if Five-Elements Music Therapy works to treat depression disorder. It will also learn about the mechanism of action of Five-Elements Music Therapy of Traditional Chinese Medicine (TCM) for depression disorder. The main questions it aims to answer is: Can Five-Elements Music Therapy, primarily using Gong-mode and Zhi-mode tones, improve Hamilton Depression Rating Scale (HAMD) scale scores in patients with depression disorder by regulating prefrontal cortex function?

Researchers will compare customized five-element music 1 (featuring Gong-mode and Zhi-mode as the predominant tones) to customized five-element music 2 (featuring Shang-mode and Yu-mode as the predominant tones, with identical rhythm and pitch to music 1), while simultaneously observing electroencephalogram (EEG), eye movement, and pulse diagnostic data from a healthy control group, to see if customized five-element music 1 featuring Gong-mode and Zhi-mode as the predominant tones can significantly improve depressive states in patients with depressive disorder.

Participants will:

1. Undergo Five-Element Music 1 or Five-Element Music 2 therapy twice daily for 4 weeks (28 days), with each session consisting of 30 minutes of music listening followed by 10 minutes of rest.
2. Concurrently receive antidepressant therapy with fluoxetine hydrochloride.
3. Undergo relevant examinations once every two weeks and record their levels of depression and anxiety (Hamilton Depression Rating Scale (HAMD) & Hamilton Anxiety Rating Scale (HAMA)).
4. Undergo and record their post-intervention electroencephalogram (EEG), eye movement, and pulse characteristics after the 4-week period.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for depressive episodes of ICD-10;
* Hamilton Depression Scale -17 items score ≥14 points;
* The diagnosis should be confirmed by at least two physicians with the title of attending physician or above.
* Have sufficient visual and auditory levels to ensure that the necessary checks and experiments for the research can be completed;
* Sign the written informed consent form and agree to be enrolled in the trial as required by the research plan.

Exclusion Criteria:

* There are serious heart, liver and kidney diseases, organic brain diseases, serious cardiovascular diseases, tumors, blood history, rheumatism, malnutrition and neurodegenerative diseases, etc.
* Depressive episodes secondary to other mental or physical illnesses;
* There is a history of abuse of tobacco, alcohol and other psychoactive substances;
* Those with comorbidities of other mental disorders;
* Had participated in other drug clinical trials before inclusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The reduction rate of Hamilton Depression Rating Scale-17（HAMD-17） after treatment | From enrollment to the end of the treatment at 4 weeks
  Reduction rate = (Baseline HAMD-17 score - Week 4 HAMD-17 score) / Baseline HAMD-17 score. A HAMD-17 response rate ≥50% is defined as an effective treatment

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale（HAMA） | From enrollment to the end of treatment at 4 weeks
  HAMA scale is used to assess the severity of anxiety symptoms in patients with neurotic disorders and other conditions. Previous studies have reported good reliability and validity for this scale. According to the evaluation criteria provided by the Chinese Psychiatric Rating Scale Cooperative Group:
  1. A total score above 29 indicates severe anxiety;
  2. Above 21 indicates definite marked anxiety;
  3. Above 14 indicates definite anxiety;
  4. Above 7 suggests possible anxiety;
  5. Below 7 signifies no anxiety symptoms. Previous studies have commonly used 14 as the cut-off score, with higher total scores indicating more severe anxiety symptoms.
Repeatable Battery for the Assessment of Neuropsychological Status（RBANS） | From enrollment to the end of treatment at 4 weeks
  This scale is used to assess participants' cognitive function. It offers advantages in clinical applications including concise administration, user-friendly operation, and sensitive/responsive results. Patients experiencing depressive episodes demonstrate high compliance with completion. The RBANS includes five domain scores:
  * Immediate Memory: Reflects the participant's ability to retain information immediately after presentation;
    * Visuospatial/Constructional: Reflects the participant's ability to perceive spatial relationships and accurately reproduce drawings;
      * Language: Reflects the participant's verbal fluency and naming abilities; ④ Attention: Reflects the participant's working memory capacity and ability to access short-term memory stores through visual and verbal modalities; ⑤ Delayed Memory: Reflects the participant's anterograde memory capacity.
Treatment Emergent Symptom Scale（TESS） | From enrollment to the end of treatment at 4 weeks
  Among comparable scales, it provides the most comprehensive item coverage-assessing both common adverse symptoms/signs and multiple laboratory findings. The Treatment Emergent Symptom Scale (TESS) requires clinicians to evaluate each symptom across three dimensions: Severity, Relationship to Intervention, and Action Taken.
  Severity is rated on a 0-4 scale:
  0 = Absence of the symptom;
  1. = Occasional presence of the symptom;
  2. = Mild severity, no impairment to routine functioning;
  3. = Moderate severity, producing some impairment to routine functioning;
  4. = Severe, causing significant impairment or disability to routine functioning.
Event-related potential（ERP） | From enrollment to the end of treatment at 4 weeks
  ERP data acquisition in the laboratory was performed using the Curry system with an internationally standard 64-channel electrode cap. The right mastoid (M2) served as the reference electrode. Electrodes were attached above and below the left orbit to record vertical electro-oculogram (VEOG), and electrodes were placed at the outer canthi of both eyes to record horizontal electro-oculogram (HEOG). ERP data acquisition commenced once all electrode impedances were reduced below 5 kΩ.
  For ERP data analysis, the recorded signals were band-pass filtered between 0.1 Hz and 30 Hz and continuously sampled at 500 Hz. The data were segmented into epochs of 1700 ms duration, including a 200-ms pre-stimulus baseline period and a 1500-ms post-stimulus period. The peak amplitudes of ERP components were calculated separately for each experimental group.
Eye Movement（EM） | From enrollment to the end of treatment at 4 weeks
  Participant Preparation: Adjust the chair height and chin rest so that the participant's horizontal line of sight aligns with the center of the screen or the center of the upper half of the screen. Adjust the orientation of the eye tracker using its mount to ensure the eye being tracked is centered in the image on the operator's monitor.
  Calibration: Perform calibration using the eye tracker to ensure the participant's eye is within its field of view. Ensure accurate identification of the eye and corneal reflection points through automatic threshold adjustment or manual adjustment. Instruct the participant to fixate on calibration points displayed on the screen to begin the calibration process.
  Data Recording: Once calibration is successful, begin presenting the stimulus materials and recording the data.
  Data Saving: Upon completion of the experiment, the data will be automatically saved to the designated folder.
Pulse diagnosis data | From enrollment to the end of treatment at 4 weeks
  Participant Preparation: Ensure the participant is seated comfortably with their arm extended level with the heart, wrist straight, palm facing upwards. Place a fabric cushion under the wrist joint (dorsal side).
  Device Connection: A Traditional Chinese Medicine (TCM) practitioner determines the Guan pulse position. Connect the sensor to this location.
  Data Recording: The operator uses the software to record the participant's pulse pattern in a resting state. A typical recording duration is 1 minute.
  Data Saving: Upon completion of the experiment, the data will be automatically saved to the designated folder.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT07048938/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent Form for Participants (Intervention Group) (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT07048938/ICF_001.pdf
  • Informed Consent Form: Informed Consent Form for Participants (Healthy Group) (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT07048938/ICF_002.pdf